CLINICAL TRIAL: NCT00549744
Title: A Randomized, Double-blind, Double-dummy, Placebocontrolled,Three-period, Incomplete Block, Crossover Study, to a Investigate the Effect of 14 Days Repeat Inhaled Dosing With GSK256066 in Mild/Moderate Asthmatic Patients.
Brief Title: Clinical Endpoint Trial Investigating Once Daily and Bronchodilator Dosing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: IPA107948
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: ASTHMA; CLINICAL ENDPOINT,
MeSH Terms: conditions — Asthma | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256066

SUMMARY:
Subjects will attend the unit for out-patient visits on Day 1, Day 7, Day 14 and Day 15 of each treatment period. The washout period between each treatment period will be a minimum of 10 days and maximum of 28 days. Subjects will participate in 3 treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinically stable persistent mild/moderate asthma within the 4 weeks preceding the screening visit, with the exclusion of other significant pulmonary diseases (e.g. chronic bronchitis, emphysema, bronchiectasis, cystic fibrosis or bronchopulmonary dysplasia)
* Subjects with a screening pre-bronchodilator FEV1 70% predicted (having abstained from bronchodilators for the required period). Predicted values are based on the NHanes normal ranges
* During the screening visit, subjects must demonstrate the presence of reversible airway disease, defined as an increase in FEV1 of 12.0% over the max of the three screening measures and an absolute change of 150 mL within 30 minutes following a single 400 mg salbutamol dose
* Male and females who are aged between 18 and 65 years of age.A female is eligible to enter and participate in the study if she is of:

  1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who is post menopausal. For the purposes of this study, post menopausal is defined as 1 year without menses (FSH/LH will be also tested to confirm menopausal status); or
  2. Child bearing potential, has a negative pregnancy test (urine) at screening and pre-dose Day 1, and agrees to one of the following acceptable contraceptive methods when used consistently and correctly (i.e., in accordance with the approved product label and the instructions of a physician for the duration of the study - screening visit to follow-up contact):

Complete abstinence from intercourse from the screening visit, throughout the trial and for 7 (~5 half-lives of GSK256066) days after the completion of the trial; or Male partner was sterile prior to the female subject's entry into the study, or Implants of levonorgestrel inserted for at least 1 month prior to the study medication administration but not beyond the third successive year following insertion; or Injectable progestogen administered for at least 1 month prior to the study medication administration and administered for 1 month following study completion; or Oral contraceptive (combined or progestogen only) administered for a least one monthly cycle prior to study medication administration; or The contraceptive transdermal patch, Ortho Evra (if the subject is less than 89kg); or Double-barrier method - spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a spermicide and female diaphragm.

Recent data now shows that certain double-barrier methods have a failure rate below 1% [Trussell, 2003]. Specifically, these are a spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a female diaphragm). This provides validated confirmation of the failure rate of the double-barrier method. Thus this method now meets the stated criterion for acceptable contraception in the EMEA guidelines [CPMP/ICH/285/95, 2000]; or Condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; or An intrauterine device (IUD) or intrauterine system (IUS), inserted by a qualified physician, with published data showing that the highest expected failure rate is less than 1% per year; (not all IUDs meet this criterion) Acceptable IUDs: Tcu-380A (Paragard), TCU-380 Slimline (Gyne T Slimline), Tcu-220C, MULTILOAD-250 (MLCu-250) and 375, NOVA T and CUNOVAT (Novagard), Levonorgesterol (LNG-20) Intra-uterine System (Mirena/Levonova), and FlexiGard 330/CuFix PP330 (Gynefix). The device must be inserted at least 2 weeks prior to the Screen visit, and remain throughout the study and through the follow-up phase of the study or Any other methods with published data showing that the highest expected failure rate is less than 1% per year.

* Body weight of 50 kg and Body mass index within range of 19-31 kg/m2 inclusive
* Subjects who are current non-smokers, who have not used any inhaled tobacco products (snuff is permitted) in the 12 month period preceding the screening visit and who have a pack history of £ 10 pack years
* No significant abnormality on 12-lead ECG at screening, including the following requirements:

Ventricular rate ≥ 40 beats per minute PR interval ≤ 200 ms Q waves < 30 ms (up to 50 ms permitted in lead III only) QRS interval to be ≥ 60 ms and ≤ 110 ms QTc interval < 450msec (QTcB or QTcF; machine or manual reading) based on a single ECG value, or an average from three ECGs obtained over a brief recording period

* Able to provide written informed consent
* The subject is able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions
* Demonstrated ability to use the inhaler device in a satisfactory and repeatable manner

Exclusion Criteria:

* As a result of medical interview, physical examination or screening investigations, the principle investigator or delegate physician deems the subject unsuitable for the study. Subjects must not have a systolic blood pressure above 145 mmHg or a diastolic pressure above 85 mmHg unless the Investigator confirms that it is satisfactory for their age
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease*, haematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, bronchiectasis or pulmonary fibrosis)
* Subjects will require normal serum creatinine clearance values at screening [calculated from serum creatinine by a predicting equation using Cockcroft-Gualt formula]. If the creatinine clearance value is greater than the upper limit of normal as determined by the local laboratory reference range, the Investigator will determine whether this is a clinically significant finding that would preclude participation
* Subject has a history of atrial arrhythmia or ventricular arrhythmia
* Pregnant or nursing females
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception from at least two weeks prior to the first dose of study medication; and to continue until the final pregnancy test has been performed (not less than 150 hours after treatment
* Subjects with a history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with either respiratory arrest or hypoxic seizures
* Asthma exacerbations requiring treatment with oral corticosteroids: any exacerbations within 3 months of the screening visit or two or more exacerbations within 6 months of the screening visit or admittance to hospital for an asthma exacerbation within 1 year of the screening visit
* Subjects who have suffered an upper or lower respiratory tract infection within 4 weeks of the screening visit
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* Subjects who are unable to washout the following protocol defined prohibited medications within the defined times at screening:

Oral corticosteroids Inhaled, intranasal and topical steroids Long acting beta agonists Short acting beta agonists

* The subject has taken prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is the longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety
* History of alcohol/drug abuse or dependence within 12 months of the study
* Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine)
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Donation of blood in excess of 500 mL within a 56 day period prior to dosing
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* The subject has tested positive for HIV antibodies (if tested according to site SOPs)
* The subject has a positive pre-study urine drug/ urine alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-11-16 (Actual); Primary Completion 2008-08-27 (Actual); Study Completion 2008-08-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (pre-bronchodilator and pre-dose) forced expiratory volume at 1 second (FEV1) on Day 14 | Baseline (Day 1, pre-dose) and Day 14 of each treatment period
  FEV1 is a lung function measure defined as the maximal amount of air that can be forcefully exhaled in one second. Mean FEV1 from the 3 acceptable spirometric efforts were recorded after withholding salbutamol used as bronchodilator at all visits for at least 6 hours (h) and at pre-dose. Baseline was defined as the mean of the 3 pre-dose measurements on Day 1 of each treatment period. The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (pre-dose, Day 14) value. Adjusted mean was reported as least square (LS) mean.

SECONDARY OUTCOMES:
Change from Baseline (pre-bronchodilator and pre-dose) FEV1 on Day 7 and at one h post-dose on Day 7 and Day 14 | Day 1 (Baseline, pre-dose), Day 7 and Day 14 of each treatment period
  FEV1 is a lung function measure defined as the maximal amount of air that can be forcefully exhaled in one second. Mean FEV1 from the 3 acceptable spirometric efforts were recorded after withholding salbutamol used as bronchodilator at all visits for at least 6 h and at pre-dose on Day 7, one h post-dose on Day 7 and one h post-dose on Day 14. Baseline was defined as the mean of the 3 pre-dose measurements on Day 1 of each treatment period. The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (pre-dose Day 7, one h post-dose on Day 7 and one h post-dose on Day 14) values. Adjusted mean was reported as LS mean.
Change from Baseline in FEV1 over 12 h post-dose on Day 1 | Baseline (Day 1, pre-dose) and Day 1 (0.5 h, 1 h, 2 h, 8 h and 12 h post-dose) of each treatment period
  FEV1 is a lung function measure defined as the maximal amount of air that can be forcefully exhaled in one second. Mean FEV1 from the 3 acceptable spirometric efforts were recorded after at pre-dose, 0.5 h, 1 h, 2 h, 8 h and 12 h post-dose on Day 1. Baseline was defined as the mean of the 3 pre-dose measurements on Day 1 of each treatment period. The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (0.5 h, 1 h, 2 h, 8 h and 12 h post-dose) values on Day 1. Adjusted mean was reported as LS mean.
Change from Baseline in FEV1 over 12 h post-dose on Day 14 | Baseline (Day 1, pre-dose) and Day 14 (0.5 h, 1 h, 2 h, 8 h and 12 h post-dose) of each treatment period
  FEV1 is a lung function measure defined as the maximal amount of air that can be forcefully exhaled in one second. Mean FEV1 from the 3 acceptable spirometric efforts were recorded after at pre-dose, 0.5 h, 1 h, 2 h, 8 h and 12 h post-dose on Day 1. Baseline was defined as the mean of the 3 pre-dose measurements on Day 1 of each treatment period. The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (0.5 h, 1 h, 2 h, 8 h and 12 h post-dose) values on Day 14. Adjusted mean was reported as LS mean.
Mean change from Baseline (pre-bronchodilator and pre-dose) Peak Expiratory Flow Rate (PEFR) averaged over the 14-day period | Baseline (Screening, 7 days prior to Day 1 of Treatment period 1) and Day 1 to 14 of each treatment period
  PEF is a measure of lung function and measures how fast a person can breathe out. It was measured using a peak flow meter by the participants and recorded on diary cards during Day 1 to Day 14 pre-dose am and pm of each treatment period. The efforts were recorded after withholding salbutamol used as bronchodilator for at least 6 hours. The averaged PEFR over the 14-day treatment period was calculated as the mean of the 14 pre-dose observations during each treatment period. Baseline was defined as the assessment done during Screening (the average of am and average of pm measurements over the last 7 days pre-dose prior to Day 1 of treatment period 1). The change from Baseline was calculated by subtracting the Baseline value (average of am and average of pm screening values) from the individual post-Baseline (average of am and average of pm values over 14 days) values. Adjusted mean was reported as LS mean.
Mean change from Baseline ratio of exhaled nitric oxide on Day 1, Day 7 and Day 14 | Baseline (Day 1 pre-dose), Day 7 and Day 14 of each treatment period
  The exhaled nitric oxide assessment is used as a marker for airway inflammation. The exhaled nitric oxide was assessed using breath test on Day 1 (pre-dose and 1 h post-dose on Day 1), Day 7 (pre-dose) and Day 14 (pre-dose, 1 h and 24 h post-dose). Baseline was defined as the assessment done pre-dose on Day 1. The change from Baseline was calculated by subtracting the Baseline value (Day 1, pre-dose) from the individual post-Baseline (1 h post-dose Day 1, pre-dose Day 7 and Day 14 at pre-dose, 1 h post-dose and 24 h post-dose) values. Data was analyzed using repeated measures mixed effects model for the ratio of change from Baseline values, derived from dividing doses of GSK256066 by placebo, adjusted for period, treatment, Day (1, 7 or 14), time (pre-dose, 1 or 24 h), period-level Baseline of exhaled nitric oxide and participant-level Baseline exhaled nitric oxide as fixed effects and participant as a random effect. Adjusted geometric mean is reported as LS geometric mean.
Mean provocative concentration of methacholine resulting in a 20% reduction in FEV1 (PC20) on Day 15 | Day 15 of each treatment period
  The PC20 was assessed using the methacholine challenge. This is a physiological measurement derived from repeated breathing maneuvers which measures airway reactivity. Participants were exposed to higher and higher concentrations of an airway irritant (in this case methacholine), and between each dose spirometry was performed. The test was stopped after the FEV1 fell 20% below the Baseline. The concentration of methacholine at which this occurred was called the PC20. The methacholine challenge was performed at 24 h post-dose on Day 14 (morning of Day 15) after exhaled nitric oxide assessment. Data was analyzed using mixed effect model, where the model was adjusted for period and treatment as fixed effects and participant as a random effect. Adjusted geometric mean is reported as LS geometric mean.
Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC [0-t]) and to infinity (AUC [0-infinity]) of GSK256066 at Day 1 and Day 14 | Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h)
  Blood samples were collected on Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h). The AUC (0-t) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. AUC (0-infinity) was planned to be calculated, where data permitted, as the sum of AUC (0-t) and Ct/z, where Ct was the observed plasma concentration obtained from the log-linear regression analysis of the last quantifiable time-point and z is the terminal phase rate constant. Data for AUC (0-infinity) was not derived due to non quantifiable data.
Maximum observed concentration (Cmax) of GSK256066 at Day 1 and 14 | Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h)
  Blood samples were collected on Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h). The first occurrence of the Cmax was determined directly from the raw concentration-time data.
Time of occurrence of Cmax (Tmax) and time to apparent terminal elimination phase half-life (t1/2) of GSK256066 at Day 1 and Day 14 | Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h)
  Blood samples were collected on Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h). The time at which Cmax was observed was determined directly from the raw concentration-time data. The t1/2 was planned to be obtained as the ratio of ln2/λz, where λz is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data. The data for t1/2 was not derived due to non quantifiable data.
AUC (0-t) and AUC (0-infinity) of GSK614917 at Day 1 and Day 14 | Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h)
  GSK614917 is a metabolite of GSK256066. Blood samples for PK analysis were collected on Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h). The AUC 0-t was planned to be determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. AUC (0-infinity) was planned to be calculated, where data permitted, as the sum of AUC (0-t) and Ct/z, where Ct was the observed plasma concentration obtained from the log-linear regression analysis of the last quantifiable time-point and z is the terminal phase rate constant. Data for this outcome measure was not derived due to non quantifiable data.
Cmax of GSK614917 at Day 1 and Day 14 | Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h)
  GSK614917 is a metabolite of GSK256066. Blood samples for PK analysis were collected on Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h). The first occurrence of the Cmax was planned to be determined directly from the raw concentration-time data. Data for this outcome measure was not derived due to non quantifiable data.
Tmax and t1/2 of GSK614917 at Day 1 and Day 14 | Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h)
  Blood samples were collected on Day 1 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h and 12 h) and Day 14 (pre-dose, 0.25 h, 0.5 h, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h and 24 h). The time at which Cmax was observed was planned to be determined directly from the raw concentration-time data. The t1/2 was planned to be obtained as the ratio of ln2/λz, where λz is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data. Data for this outcome measure was not derived due to non quantifiable data.
Number of participants with any adverse event (AE), serious adverse event (SAE) or death | Up to Follow-up (18 weeks)
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Number of participants with abnormal both clinically non-significant (CNS) and clinically significant (CS) electrocardiograph (ECG) values | Up to Day 14 of each treatment period
  The ECG measurements were made with the participant in a supine position having rested in this position for at least 10 minutes before each time-point. 12-lead ECG assessments were obtained on Day 1 (pre-dose triplicate assessment, 0.5 h, 1 h, 2 h, 8 h and 12 h), Day 7 (pre-dose) and Day 14 (pre-dose, 0.5 h, 1 h, 2 h, 8 h, 12 h and 24 h) using a machine that automatically calculated PR, QRS, QT and QTcB. Abnormal ECG findings (CNS and CS) were categorized. The abnormal PCI range included QTc interval of <300 and >500 milliseconds (msec) and increase from baseline QTc interval of >60 msec, PR interval <110 and >220 msec and QRS interval <75 and >110 msec. Baseline was Day 1 (mean of triplicate assessments done at pre dose).
Number of participants with hematology abnormalities of potential clinical importance (PCI) during the treatment period | Up to Day 14 of each treatment period
  The assessments were done at pre-dose on Day 1, Day 7 and Day 14 of each treatment period. The following laboratory parameters of clinical haematology were analyzed: platelet count, red blood cells (RBC) count, absolute white blood cells (WBC) count, reticulocyte count, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), total neutrophils, lymphocytes, monocytes, eosinophils and basophils. Only those parameters for which at least one value of PCI was reported are summarized.
Number of participants with clinical chemistry abnormalities of PCI during the treatment period | Up to Day 14 of each treatment period
  The assessments were done at pre-dose on Day 1, Day 7 and Day 14 of each treatment period. The following laboratory parameters of clinical chemistry were analyzed: blood urea nitrogen (BUN), creatinine, total cholesterol, sodium, potassium, chloride, total bicarbonate, calcium, C-reactive protein (CRP), aspartate aminotransferase (AST), alanine amino transferase (ALT), gamma glutamyltransferase (GGT), alkaline phosphatase, creatine kinase (CK), lactate dehydrogenase (LDH), total and direct bilirubin, uric acid, albumin and total protein. Only those parameters for which at least one value of PCI was reported are summarized.
Number of participants with abnormal urinalysis results | Up to Day 14 of each treatment period
  The assessments were done at Day 1, Day 7 and Day 14 for urine glucose, protein, occult blood, ketones, nitrites, bilirubin, leukocytes esterase and urobilinogen by dipstick. The participants were categorized with results of 1 +, 2+, 3+, 4+, 7+, positive, trace, not rated (NR), 0, 0.2, 1, 16 and 3.2. Only those parameters for which at least one value of these categories reported are summarized.
Number of participants with vital sign value of PCI during the treatment period | Up to Day 14 of each treatment period
  The assessments were done at pre-dose on Day 1 (taken in triplicate at pre-dose, 0.5, 1, 2, 8 and 12 h post-dose), Day 7 (pre-dose) and Day 14 (24 h post-dose) of each treatment period. Supine vital signs measurements were made with the participant in a supine position having rested in that position for at least 5 minutes before the first reading at each time point. Vital signs assessment included heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP). Criteria for vital sign values meeting PCI included: SBP < 70 millimeters of mercury (mmHg) and > 160 mmHg; DBP < 45 mmHg and > 110 mmHg; < 35 beats per minute and > 160 beats per minute. Only those parameters for which at least one value of PCI was reported are summarized.
Number of participants with troponin results | Up to Day 14 of each treatment period
  The assessment of troponin (I and or T) was done to ensure participants safety and further characterize potential renal and cardiac effects. It was monitored at pre dose on Day 1, Day 7 and Day 14. Data is categorized according to the troponin levels of <0.03 µg/L, >0.03 µg/L but <0.10 µg/L and negative. The PCI value for troponin T: low= 0 µg/L and high >0.4 µg/L.
Genetic variations of participants for relationship between genetic variants and or PK, tolerability and efficacy of GSK256066 | At any time post-Randomization
  This included the study of variability in drug response due to hereditary factors in different populations. There is increasing evidence that an individual's genetic composition (i.e., genotype) may impact the pharmacokinetics (absorption, distribution, metabolism, elimination), pharmacodynamics (relationship between concentrations and pharmacologic effects or the time course of pharmacologic effects) and/or clinical outcome (in terms of efficacy and/or safety and tolerability). A whole blood sample (10ml) was planned to be collected. The data for this outcome measure was not collected.
Mean phosphodiesterase-4 (PDE4) values | Day 7 of each treatment period
  PDEs are a super family of enzymes that catalyze the breakdown of cyclic adenosine monophosphate (cAMP) and/or cyclic guanosine monophosphate (GMP) to their inactive form. PDE4 is the main selective cAMP-metabolizing enzyme in inflammatory and immune cells. Because PDE4 is highly expressed in leukocytes and other inflammatory cells involved in the pathogenesis of inflammatory lung diseases, such as asthma, inhibition of PDE4 had been predicted to have an anti inflammatory effect for them. PDE4 was assessed in sputum samples, collected 2-3 h post-dose on Day 7 by transcriptomic analysis on sputum ribonucleic acid (RNA) samples. Data is reported for PDE4B.
Mean differential cell counts during sputum analysis | Day 7 of each treatment period
  Sputum samples were collected 2-3 h post-dose on Day 7 to measure the differential cell counts which is used as an indicator of the anti-inflammatory activities. The cells include neutrophils, macrophages, lymphocytes, total leukocyte count and bronchial epithelial cells.
Biomarkers of sputum analysis | Day 7 of each treatment period
  The anti-inflammatory activity was assessed by measuring novel candidate biomarkers of the biological response associated with the action of GSK256066, in sputum samples, collected 2-3 h post-dose on Day 7 by transcriptomic analysis on sputum ribonucleic acid (RNA) samples. Data is reported for the biomarkers of glyceraldehyde-3-phosphate dehydrogenase (GAPDH), oncostatin M (OSM), cyclophilin, B actin, suppressor of cytokine signaling 3 (SOCS3), ETS proto-oncogene 2 transcription factor (ETS2), amphiregulin (AREG), cAMP responsive element modulator (CREM) and salt inducible kinase 1 (SNF1LK).
Mean interleukin-10 (IL-10), IL-13 and tumour necrosis factor alfa (TNFα) values | Day 7 of each treatment period
  Cytokine sampling was planned of Day 7, 2-3 h post-dose to measure the IL10, IL-13 and TNFα for anti-inflammatory activity in sputum. However the data was not collected for this outcome measure.
Anti inflammatory activity in sputum assessed by SNF1LK Cytospin on Day 7 | Day 7 of each treatment period
  Sputum samples were collected 2-3 h post-dose on Day 7 to measure the anti-inflammatory activities by SNF1LK nuclear intensity of staining and cytoplasmic intensity of staining of the cells.
Anti-inflammatory activity in sputum assessed by ratio of SNF1LK Cytospin on Day 7 | Day 7 of each treatment period
  Sputum samples were collected 2-3 h post-dose on Day 7 to measure the anti-inflammatory activities by the ratio of SNF1LK nuclear intensity of staining and cytoplasmic intensity of staining of the cells.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Wellington, New Zealand
- South Africa (2):
  - GSK Investigational Site, George, Eastern Cape
  - GSK Investigational Site, Bloemfontein